CLINICAL TRIAL: NCT06050928
Title: Phase 1b, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of EP262 in Subjects With Chronic Inducible Urticaria (CALM-CIndU)
Brief Title: Phase 1b, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of EP262 in Subjects With Chronic Inducible Urticaria
Acronym: CALM-CIndU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-262-102
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Chronic Inducible Urticaria
MeSH Terms: conditions — Chronic Inducible Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EP262 150 mg (Experimental): Once daily
  Interventions: Drug: Oral EP262

INTERVENTIONS:
Drug: Oral EP262 — Once daily

SUMMARY:
This phase 1b trial will evaluate the effects of EP262 in subjects with Chronic Inducible Urticaria (CIndU), including symptomatic dermographism and cold urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CIndU (symptomatic dermographism or cold urticaria) for greater than 3 months and positive response to applicable skin provocation testing
* Willing to discontinue chronic treatment with antihistamines during the study

Exclusion Criteria:

* Urticaria with a clear underlying etiology other than symptomatic dermographism or cold urticaria
* Other active skin diseases that might confound the study evaluations (eg, atopic dermatitis, bullous pemphigoid, prurigo nodularis, dermatitis herpetiformis)
* Regularly experience wheals covering the area of the body where skin testing will be conducted (eg, more than one third of the volar surface of the forearms)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EP262 | Measured from Day 1 to End of Study or Early Termination (up to 12 weeks)
  Assessed by the incidence of treatment-emergent adverse events

SECONDARY OUTCOMES:
Change in Critical Friction Threshold (CFT) | Measured from Baseline to Week 4
  Assessed by the number of prongs that elicit a wheal response using a FricTest (in subjects with symptomatic dermographism)
Change in Critical Temperature Threshold (CTT) | Measured from Baseline to Week 4
  Assessed as the highest temperature that elicits a wheal response using a TempTest (in subjects with cold urticaria)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Advanced Clinical Research Institute, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research, LLC., North Charleston, South Carolina
- Canada (2):
  - Innovaderm Research Inc., Montreal
  - Gordon Sussman Clinical Research Inc., North York
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - Institut fur Allergieforschung Charite - Universitatsmedizin Berlin, Berlin
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands
- Spain (2):
  - Hospital del Mar, Barcelona
  - Hospital Arnau de Vilanova, Valencia